CLINICAL TRIAL: NCT07115537
Title: The Prognostic Significance of Platelet to White Blood Cell Ratio (PWR) in Patients With Acute Myeloid Leukemia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaymaa Abd El-Wahab El-Sadek, residant doctor at Assiut university hospital, Assiut University
Other Study IDs: PWR Acute Myeloid Leukemia
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: patients with Acute Myeloid Leukemia

SUMMARY:
Acute Myeloid Leukemia (AML) is a malignant hematological disease characterized by clonal proliferation of myeloid precursors with a reduced capacity for differentiation. It leads to accumulation of immature blasts in bone marrow (BM), peripheral blood (PB), and other tissues (Döhner et al. 2017). AML is the most common type of acute leukemia in adults, with an incidence of approximately 4 cases per 100,000 individuals per year. It predominantly affects older adults with a median age at diagnosis of 68 years (Siegel et al. 2023).

The etiology of AML is complex and multifactorial, involving genetic mutations, chromosomal abnormalities, environmental exposures, and pre-existing hematological conditions such as myelodysplastic syndromes (MDS) (Papaemmanuil et al. 2016). Advances in genomic profiling have revealed that mutations in genes such as FLT3, NPM1, IDH1/2, and TP53 play a critical role in the pathogenesis and prognosis of AML (Döhner et al. 2022).

In recent years, there has been a growing interest in using systemic inflammatory markers derived from complete blood counts (CBC) as valuable and cost-effective prognostic indicators. Ratios such as the neutrophil-to-lymphocyte ratio (NLR), plateletto- lymphocyte ratio (PLR), and lymphocyte-to-monocyte ratio (LMR have shown prognostic value in various cancers, including AML (Zhang et al. 2021). Platelets have been recognized not only for their hemostatic role but also for their involvement in tumor biology, immune modulation, and inflammation. Conversely, elevated white blood cell (WBC) counts in AML often represent a high leukemic burden and are associated with worse clinical outcomes (Döhner et al. 2015; Arber et al. 2016).

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* both sex
* Patients with Acute Myeloid Leukemia

Exclusion Criteria:

* patients with other hematological diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Acute Myeloid Leukemia
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
accuracy of Platelet to White Blood Cell Ratio (PWR) | baseline
  The accuracy of Prognostic Significance of Platelet to White Blood Cell Ratio (PWR) in Patients with Acute Myeloid Leukemia